CLINICAL TRIAL: NCT02223962
Title: The Effects of a Physical Activity Counseling Program Immediately After an Exacerbation in Patients With COPD.
Brief Title: Effects of Physical Activity Counseling After an Exacerbation in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Marc Decramer, Prof. Dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S55086; ML8991 (Other: University Hospital Leuven)
Record Dates: First submitted 2013-09-04; First posted 2014-08-22 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: COPD Exacerbation
Keywords: physical activity; COPD; activity monitors
MeSH Terms: conditions — Motor Activity; Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity (Experimental): The fitbit Ultra was used to provide real-time feedback on physical activity. An experienced physiotherapist contacted the subjects 3 times a week to receive information about the amount of steps from the previous days. In agreement with the patient, a new goal for the coming weeks was set and patients were motivated to achieve their individual goal.
  Interventions: Behavioral: Physical activity
- Usual Care (Placebo Comparator): During the hospital stay, the patients in the control group will be informed about the beneficial effects of being physically inactive.They will not receive feedback about their activities performed and will not be stimulated to become more active.
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — Counseling about physical activity will only be provided in the intervention group by 3 weekly telephone contacts. Based on the information the physiotherapist receives, he or she will adapt the goal (in agreement with the patient) and motivate the patient to reach the individual goal.

SUMMARY:
Severe exacerbations are prevalent in a subgroup of patients with COPD and generally warrant a hospitalization. During the hospitalization, patients are extremely physically inactive with only a limited recovery one month after discharge. Physical inactivity is associated with negative health benefits. Therefore intervening in the period after and exacerbation seems useful to improve the levels of physical activity. Physical activity counseling and real-time feedback have already been applied in stable patients with COPD, with beneficial effects.The present study will investigate whether this specific intervention will help to improve the activity level in patients after an acute exacerbation. Further we investigated the effects of the intervention on improvements in functional exercise capacity.

DETAILED DESCRIPTION:
After signing the informed consent, the patients will be randomized into a control group, receiving usual care, or the intervention group receiving real-time feedback and physical activity counseling.

Intervention: Physical activity counseling will be provided by 3 weekly telephone contacts based on the step count from the Fitbit Ultra. In agreement with the patient and based on the step counts a patients provided, a new goal for the next week was set. The goal was to strive for the highest possible level of physical activity during one month.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Chronic Obstructive Lung Disease (Tiff<70%)
* Hospitalized because of exacerbation
* Capable of working with electronic devices

Exclusion Criteria:

* Orthopedic/Neurologic problems making it difficult to be active
* Participation in a rehabilitation program

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Improvement in physical activity | 1 month
  The Dynaport MoveMonitor, a valid device in patients with COPD, was used to accurately measure the level of physical activity. The device was provided 3 times to the patients (baseline, after 2 weeks, after 1 month). The amount of steps, measured by this device, was used as the outcome measure.

SECONDARY OUTCOMES:
Improvement in functional exercise capacity | 1 month
  Functional exercise capacity was measured by the six minutes walking distance test (6MWD; meter). This measurement was performed at baseline and after 1 month.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Hornikx M, Demeyer H, Camillo CA, Janssens W, Troosters T. The effects of a physical activity counseling program after an exacerbation in patients with Chronic Obstructive Pulmonary Disease: a randomized controlled pilot study. BMC Pulm Med. 2015 Nov 4;15:136. doi: 10.1186/s12890-015-0126-8. PMID 26530543